CLINICAL TRIAL: NCT03436459
Title: Comparative Study of Shock Wave Therapy and Low Level Laser Therapy Effect in Patients With Myofascial Pain Syndrome of the Trapezius
Brief Title: Effects of Extracorporeal Shock Wave Therapy and Low Level Laser Therapy in Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petz Aladar County Teaching Hospital (Other)
Responsible Party: Principal Investigator, Márta Király, chief physician, Petz Aladar County Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PetzAladarCTH
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Myofascial Pain Syndrome
Keywords: extracorporeal shock wave therapy (ESWT); Low level laser therapy (LLLT); Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Extracorporeal Shockwave Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracorporeal shock wave therapy group (Active Comparator): Patients in the shock wave therapy group received total of 1000 shock waves for each treatment at the frequency of 10Hz, with 2 Bar pressure and energy flux density (EFD) of 0.25 mJ/mm2 per minute by using BTL-6000 SWT Topline Power® 3 times with a week's interval between the treatments.
  Interventions: Device: Extracorporeal Shock Wave Therapy
- Low Level Laser Therapy group (Active Comparator): Patients in the laser therapy group received LLLT once a day for three weeks (altogether 15 working days) to the trigger points and around them in the upper trapezius. The type of laser used: PR999 4 Watt (W) scanning laser; Medical Italia®, around trigger points with 3 Joule /centimeter² (J/cm²), power 800 milliwatt (mW), frequency 2000 Hertz (Hz), on trigger points with 9 J/cm², power 2000mW, frequency 5000Hz for total of 2 minutes on each spot.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — shock wave therapy once a week for three weeks, total of 1000 shock waves for each treatment at the frequency of 10Hz, with 2 Bar pressure and energy flux density (EFD) of 0.25 mJ/mm2 per minute using a BTL-6000 SWT Topline Power® device
  Arms: Extracorporeal shock wave therapy group
Device: Low Level Laser Therapy — LLLT once a day for three weeks (altogether 15 working days) using a PR999 4W scanning laser device; around trigger points with 3 J/cm2, power 800 mW, frequency 2000Hz, on trigger points with 9 J/cm², power 2000mW, frequency 5000Hz for total of 2 minutes on each spot
  Arms: Low Level Laser Therapy group

SUMMARY:
This study evaluates the effects of low level laser therapy and extracorporeal shock wave therapy in patients with myofascial pain syndrome of the upper trapezius. Half of the patients receive laser therapy, half of them receive shock wave therapy for three weeks.

DETAILED DESCRIPTION:
Low Level Laser Therapy (LLLT) inducing photochemical and photothermal effect, increases blood flow and vascular permeability and improves cell metabolism. All these lead to muscle recovery. It also activates somatosensory receptors of the skin and reduces local pain and muscle spasm.

The specific mechanisms of extracorporeal shock wave therapy (ESWT) in treating musculoskeletal pain remain unclear. It reduces pain and inflammation by modulating nitrogen-monoxide (NO) and vascular endothelial growth factor (VEGF). It can destroy sensory unmyelinated nerve fibers, and stimulate neovascularization and collagen synthesis in degenerative tissues.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age with myofascial pain syndrome meeting the Simon's diagnostic criteria (5 major and 1 minor) for at least 8 weeks (chronic pain)
* no physiotherapy or local injection within 3 months before starting the study

Exclusion Criteria:

* acute onset of neck pain
* physiotherapy or local injection within 3 months before starting the study
* abnormal lab test (ESR, hematology)
* infection, fever
* cervical radiculopathy
* uncontrolled hypertension, anticoagulation or defect in blood coagulation
* previous cervical operaton

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
change in severity of pain at rest | week 0 and week
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in severity of pain at rest | week 0 and week 15
  change from baseline severity of pain at rest recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in severity of pressure pain | week 0 and week 3
  change from baseline severity of pressure pain recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in severity of pressure pain | week 0 and week 15
  change from baseline severity of pressure pain recorded on a 100 mm visual analogue scale, where 0 mm represents no pain, 100 mm represents unbearable pain.
change in function (percentage of disability) | week 0 and week 3
  change from baseline Neck Disability Index (NDI) at week 3. It includes 10 part; pain intensity, personal care, lifting objects, reading, headache, concentration, work, driving, sleeping and entertainments. There are six presumptions; the first is given 0 and the last presumption has the score of 5. The total maximum score is 50, that represents 100% disability. The lower score represents better outcome.
change in function (percentage of disability) | week 0 and week 15
  change from baseline Neck Disability Index (NDI) at week 15. It includes 10 part; pain intensity, personal care, lifting objects, reading, headache, concentration, work, driving, sleeping and entertainments. There are six presumptions; the first is given 0 and the last presumption has the score of 5. The total maximum score is 50, that represents 100% disability. The lower score represents better outcome.
change in quality of life | week 0 and week 3
  change from baseline quality of life (36-Item Short Form Health Survey /SF-36/) at week 3. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more the disability, i.e. a score of zero is equivalent to maximum disability.
change in quality of life | week 0 and week 15
  change from baseline quality of life (SF-36) at week 15. It consists of eight scaled scores (vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more the disability, i.e. a score of zero is equivalent to maximum disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Petz Aladár County Teaching Hospital, Győr, Hungary

REFERENCES:
- [Derived] Kiraly M, Bender T, Hodosi K. Comparative study of shockwave therapy and low-level laser therapy effects in patients with myofascial pain syndrome of the trapezius. Rheumatol Int. 2018 Nov;38(11):2045-2052. doi: 10.1007/s00296-018-4134-x. Epub 2018 Aug 31. PMID 30171341